CLINICAL TRIAL: NCT01246778
Title: The Influence of Sunitinib on Contractility of Human Atrial Trabeculae
Brief Title: Sunitinib and Atrial Trabeculae Contractility
Acronym: SCAR
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, G. Rongen, Prof. dr. Rongen, Radboud University Medical Center
Other Study IDs: SCAR
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Cardiotoxicity; Ischemia; Heart Failure
MeSH Terms: conditions — Cardiotoxicity; Ischemia; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: None Retained — Atrial tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With/without sunitinib: Two trabeculas will be isolated and one will be exposed to sunitinib and the other to normal buffer solution. Both will be stimulated to contraction during 200 minutes.
- With/without sunitinib IP: Two trabeculas will be isolated and one will be exposed to sunitinib and the other to normal buffer solution. Both will be stimulated to contraction and ischemia/reperfusion

SUMMARY:
Rationale:

Recently, sunitinib (a tyrosine kinase inhibitor that is used for treatment of metastatic renal carcinoma and gastrointestinal stroma tumors) has been associated with development of heart failure, possibly by off-target inhibition of AMP-protein kinase. The investigators hypothesize that sunitinib reduces the contractile ability of myocardium and the tolerance against ischemia-reperfusion and that activators of AMP-protein kinase such as atorvastatin and AICAR reverse this unwanted effect of sunitinib.

Objectives:

The primary objective of the study is to investigate the effect of sunitinib on ex-vivo atrial contractile force in absence and presence of ischemia-reperfusion.

A secondary objective is to explore if atorvastatin or AICAR prevent sunitinib-induced deterioration of contractile function of human atrial trabeculas. Study design: Lab

DETAILED DESCRIPTION:
Study population: 44 (+22) patients undergoing CABG cardiac surgery with extracorporal circulation Intervention (if applicable): none (pharmacological interventions will only be performed ex-vivo in isolated atrial tissue) Main study parameters/endpoints The developed force in ex vivo atrial trabeculas during standardized stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with extracorporal circulation

Exclusion Criteria:

* Use of oral antiarrhythmics
* theophylline use
* Use of sulfonylureas
* Atrial arrythmias
* Right ventricular failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 44 patients undergoing cardiac surgery with extracorporal circulation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Force | 200 minutes
  The developed force in ex vivo atrial trabeculae during standardized stimulation.

SECONDARY OUTCOMES:
Speed | 200 minutes
  The difference in averaged maximal speed of tension reduction during relaxation between two trabeculae
Maximal Speed | 210 minutes
  The difference in averaged maximal speed of tension development during contraction between two trabeculae.

CONTACTS AND LOCATIONS:
Overall Officials: G. A. Rongen, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands